CLINICAL TRIAL: NCT03335150
Title: Cognitive Rehabilitation for Individuals With Parkinson's Disease and MCI
Brief Title: Cognitive Rehabilitation for PD
Acronym: CogSMART-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E1691-I
Record Dates: First submitted 2017-10-18; First posted 2017-11-07 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Rehabilitation; Cognition
MeSH Terms: conditions — Parkinson Disease | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Assessor are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supportive Care (Active Comparator): Support Group for PD-MCI
  Interventions: Behavioral: Supportive Care
- CogSMART-PD (Experimental): Cognitive Rehabilitation for PD-MCI
  Interventions: Behavioral: CogSMART-PD

INTERVENTIONS:
Behavioral: CogSMART-PD — Cognitive Rehabilitation for persons with PD-MCI
  Arms: CogSMART-PD
Behavioral: Supportive Care — Support Group for persons with PD-MCI
  Arms: Supportive Care

SUMMARY:
To investigate the effectiveness of a novel compensatory cognitive rehabilitation program for individuals with Parkinson's disease (PD) and mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Eligible study participants will be randomly assigned to one of two interventions: 1) Cognitive Rehabilitation (Cognitive Symptom Management and Rehabilitation Therapy for Parkinson's disease; CogSMART-PD) or 2) Supportive Care. Interventions are held within a group format consisting of approximately 5 individuals with PD. Groups will meet once per week for 1.5 hours over a 10-week period. Neuropsychological testing will be administered pre- and post-intervention as well as 6- and 12-months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease
2. Mild Cognitive Impairment
3. Over 40 years of age
4. Fluent English speaker

Exclusion Criteria:

Other neurological conditions (e.g., stroke) besides Parkinson's disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Schiehser, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care: Support Group for PD
  Supportive Care: Support Group for persons with PD
- CogSMART-PD: Cognitive Rehabilitation for PD
  CogSMART-PD: Cognitive Rehabilitation for persons with PD
Period: Overall Study
Arm/Group | Supportive Care | CogSMART-PD
Started | 55 | 55
Enrolled + Assigned Group | 54 | 55
PRE Testing Session | 53 | 55
Commenced Group | 47 | 52
POST Testing Session | 45 | 50
Completed | 45 | 50
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Care | CogSMART-PD | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.59 (7.06) | 68.22 (7.98) | 69.39 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 34 | 43 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 50 | 52 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 0 | 0
  Race: Asian | 1 | 0 | 1
  Race: Black or African American | 1 | 2 | 3
  Race: Hispanic or Latino | 2 | 3 | 5
  Race: Native Hawaiian or Pacific Islander | 1 | 1 | 2
  Race: White or Caucasian | 49 | 49 | 98
Education [Mean (Standard Deviation); unit: years] — The number of years participant received formal education
  years | 16.15 (2.41) | 15.8 (2.29) | 15.97 (2.34)
Duration of Disease [Mean (Standard Deviation); unit: months] — Time from Parkinson's disease diagnosis to enrollment Population: 54 subjects were enrolled for the Supportive Care group. 1 subject was missing the information.
  months
    number analyzed (Participants) | 53 | 55 | 108
    (all) | 69.02 (55.97) | 73.27 (45.43) | 71.18 (50.68)
Cognitive Status [Count of Participants; unit: Participants] — Cognitive status was determined using the Diagnostic Criteria for Mild Cognitive Impairment (Litvan et al., 2012). Population: 55 subjects were enrolled into the CogSMART-PD group; however, 1 participant did not meet inclusion criteria.
  Participants
    number analyzed (Participants) | 54 | 54 | 108
    Normal Cognition | 14 | 9 | 23
    Mild Cognitive Impairment | 40 | 45 | 85
Motor Symptoms [Mean (Standard Deviation); unit: seconds] — Timed Up and Go (TUG) Test, a motor assessment Population: 54 subjects were enrolled into the Supportive Care Group; however, 1 subject dropped before their baseline assessment, and 2 were unable to complete the measure in session. 55 subjects were enrolled into the CogSMART-PD group; however, 1 subject was unable to complete the measure in session.
  seconds
    number analyzed (Participants) | 51 | 54 | 105
    (all) | 12.28 (4.85) | 11.76 (3.73) | 12.01 (4.30)
Baseline Medication [Mean (Standard Deviation); unit: milligrams] — Amount of Levodopa Equivalent Dose (LED) Population: 54 subjects enrolled in the Supportive Care group; however, 1 subject's medication info was missing. 55 subjects enrolled in the CogSMART-PD group; however, 1 subject dropped before their baseline assessment.
  milligrams
    number analyzed (Participants) | 53 | 54 | 107
    (all) | 685.26 (445.71) | 764.17 (483.10) | 725.09 (464.46)

OUTCOME MEASURES:

1. Primary Outcome: Wechsler Adult Intelligence Scale-IV (WAIS-IV) Matrix Reasoning Test Total Scaled Score
Description: The WAIS-IV Matrix Reasoning test is a validated, objective measure of executive function. Scaled scores range from 0 to 26. Higher scores indicate better executive function. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: 54 enrolled in Supportive Care: 6 dropped before group started, 1 dropped before baseline, 2 dropped during group. Therefore, 45 completed measure. 55 were enrolled in CogSMART-PD: 3 dropped before group started and 2 dropped during group. Therefore, 50 completed measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 50
score on a scale | 0.22 (2.35) | 0.42 (2.43)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.6662, Mixed Models Analysis — Interaction term; Mean Difference (Final Values) = 0.4856 — Estimated Value = Standard Error (SE) of the interaction term
Statistical Analysis 2: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.1617, Mixed Models Analysis; Mean Matrix Reasoning Total (MRT) difference between two visits while controlling for intervention; Mean Difference (Final Values) = 0.2415 — estimated value = SE
Statistical Analysis 3: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.6236, Mixed Models Analysis; Mean MRT difference between two interventions while controlling for visit; Mean Difference (Final Values) = 0.5087 — estimated value = SE

2. Secondary Outcome: Delis-Kaplan Executive Functioning System (D-KEFS): 20 Questions Test Total Questions Asked Scaled Score
Description: D-KEFS: 20 Questions Test measures executive function. The range of scores is 1 - 19 with a higher score representing better executive function. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 50
score on a scale | -0.09 (2.70) | 1.06 (3.15)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.0496, Mixed Models Analysis — Interaction term; Mean Difference (Final Values) = 0.58 — Estimated value = SE of interaction term

3. Secondary Outcome: Informant Questionnaire on Cognitive Decline in the Elderly-Self Report (IQCODE-SR) Total Score
Description: The measure examines self-reported change in cognition over time. Scores range from 16 - 80, with higher scores indicating worse functioning (or more cognitive decline). Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: 54 enrolled in Supportive Care: 6 dropped before group started, 1 dropped before baseline, 2 dropped during group. Therefore, 45 completed measure. 55 were enrolled in CogSMART-PD: 3 dropped before group started, 2 dropped during group, and 1 was missing info. Therefore, 49 completed measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 49
score on a scale | -5.51 (7.84) | -8.86 (8.19)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.047, Mixed Models Analysis — Interaction term; Mean Difference (Final Values) = 1.62 — Estimated Value = SE of interaction term

4. Secondary Outcome: Cognitive Problems and Strategies Assessment (CPSA) Memory Strategies Use Score
Description: CPSA measures cognitive problems and memory strategy use. The range for scores is 0 - 90, with higher scores indicating higher frequency of using memory and thinking strategies. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: 54 enrolled in Supportive Care: 6 dropped before group started, 1 dropped before baseline, 2 dropped during group. Therefore, 45 completed measure. 55 were enrolled in CogSMART-PD: 3 dropped before group started, 2 dropped during group, and 2 were missing info. Therefore, 48 completed measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 48
score on a scale | -0.24 (11.16) | 10.17 (16.96)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.001, Mixed Models Analysis — Interaction Term; Mean Difference (Final Values) = 2.97 — Estimated Value = SE of interaction term

5. Secondary Outcome: Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) Total Score
Description: IQCODE is a self-report questionnaire for caregivers that measures possible dementia and cognitive decline of the patient. The range for scores is 26 - 130, with higher score representing worse functioning/higher cognitive decline in the patient. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: 54 enrolled in Supportive Care: 6 dropped before group started, 1 dropped before baseline, 2 dropped during group, 5 declined a caregiver, and 1 was missing info. 39 completed measure. 55 were enrolled in CogSMART-PD: 3 dropped before group started, 2 dropped during group, 2 were missing info, and 4 declined a caregiver. 44 completed measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 39 | 44
score on a scale | -4.49 (7.03) | -10.46 (12.55)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.020, Mixed Models Analysis — Interaction term; Mean Difference (Final Values) = 2.25 — Estimated Value = SE of interaction term

6. Secondary Outcome: Memory for Intention Test (MIST) Total Score
Description: MIST measures prospective memory. The range for scores is 0 - 48 with a higher score representing better prospective memory. Scores reported below are change score.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 50
score on a scale | 4 (5.43) | 2.82 (6.87)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.444, Mixed Models Analysis — Interaction term; Mean Difference (Final Values) = 1.26 — Estimated Value = SE of interaction term
Statistical Analysis 2: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.0233, Mixed Models Analysis; There is significant difference in MIST between intervention groups controlling for visit and other significant covariates; Mean Difference (Final Values) = 1.145 — estimated value = SE
Statistical Analysis 3: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p < 0.000, Mixed Models Analysis; There is significant difference in MIST between baseline and week 10 controlling for intervention group and other significant covariates; Mean Difference (Final Values) = 0.6281 — estimated value = SE

7. Secondary Outcome: World Health Organization Quality of Life (WHOQOL)-BREF Psychological Domain Transformed Score
Description: WHOQOL-BREF is a self-reported measure of quality of life. Transformed score for the psychological domain ranges from 0 to 100. Higher scores indicate better quality of life. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 49
score on a scale | 4.02 (11.60) | 0.04 (9.85)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.073, Mixed Models Analysis — Interaction term; Mean Difference (Final Values) = 2.205 — estimated value = SE of interaction term

8. Secondary Outcome: Parkinson's Disease Questionnaire-39 (PDQ-39) Total Score
Description: The PDQ-39 is a patient-reported measure of health and quality life over a 1-month period in individuals with Parkinson's disease. Total scores range from 0 to 156. Higher scores indicate poorer quality of life. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 45 | 49
score on a scale | -2.31 (11.56) | -2.69 (10.27)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.82, Mixed Models Analysis — Interaction Term; Mean Difference (Final Values) = 2.25
Statistical Analysis 2: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.0257, Mixed Models Analysis; Mean PDQ-39 difference between baseline and week 10 controlling for intervention and covariates; Mean Difference (Final Values) = 1.1172 — estimated value = SE
Statistical Analysis 3: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.1101, Mixed Models Analysis; Difference in PDQ-39 between two interventions controlling for visit and covariates; Mean Difference (Final Values) = 3.8649 — estimated value = SE

9. Secondary Outcome: Neuropsychiatric Inventory-Questionnaire (NPI-Q) Total Month Score
Description: The NPI-Q is a self-reported measure of neuropsychiatric symptoms over a 1 month period and 1 year period. Total month scores range from 0 to 156. Higher scores indicate greater severity of neuropsychiatric symptoms. Scores reported below are change scores.
Time Frame: Baseline and Week 10
Population: 54 enrolled in Supportive Care: 6 dropped before group started, 1 dropped before baseline, 2 dropped during group, 5 declined a caregiver, and 2 were missing info. 38 completed measure. 55 were enrolled in CogSMART-PD: 3 dropped before group started, 2 dropped during group, 3 were missing info, and 4 declined a caregiver. 43 completed measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care | CogSMART-PD
Number analyzed (Participants) | 38 | 43
score on a scale | 1.82 (6.63) | -2.30 (9.15)
Statistical Analysis 1: Comparison: Supportive Care vs CogSMART-PD; Test type: Other — Equality; p = 0.0263, Mixed Models Analysis — Interaction term; Median Difference (Final Values) = 1.784 — Estimated Value = SE of the interaction term

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Supportive Care | CogSMART-PD
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (N=55) | CogSMART-PD (N=55)
Clinical Motor Exam (Surgical and medical procedures) | 0 (0) | 1 (1) — Subject was surprised when neurologist administered a standard clinical motor examination to assess balance (UPDRS). As required by the exam, neurologist firmly pulled back on shoulders. Subject reported X-rays with no results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03335150/Prot_SAP_000.pdf